CLINICAL TRIAL: NCT04034758
Title: Safety and Efficacy of Heterologous Fecal Microbiota Transplantation (FMT) by Standardized Quantitative Multi-donor Intestinal Microbiota Capsule (SQIMC-md) in Mild-moderate Ulcerative Colitis Patients-a Multi-center Double-blind RCT Trial
Brief Title: Safety and Efficacy of Heterologous FMT by SQIMC-md Capsule in Mild-moderate Ulcerative Colitis Patients
Acronym: SQIMC-md
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019CR209
Record Dates: First submitted 2019-07-09; First posted 2019-07-26 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Ulcerative Colitis
Keywords: Fecal microbiota transplantation; SQIMC-md; Ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo capsule arm (Placebo Comparator): Oral administration of 30 placebo capsule containing edible pigmented starch together with full dose of oral 5-Aminosalicylic acid(5-ASA).
  Interventions: Procedure: placebo capsule
- SQIMC-md FMT arm (Active Comparator): Oral administration of 30 SQIMC-md capsules containing 2*10^13 copies of prepared fecal microbiota lyophilized powder from multiple healthy donors' fresh feces together with full dose of oral 5-Aminosalicylic acid(5-ASA).
  Interventions: Procedure: Standardized Quantitative multi-donor Intestinal Microbiota Capsule (SQIMC-md)

INTERVENTIONS:
Procedure: Standardized Quantitative multi-donor Intestinal Microbiota Capsule (SQIMC-md) — heterologous fecal microbiota transplantation (FMT) by Standardized Quantitative multi-donor Intestinal Microbiota Capsule (SQIMC-md)
  Arms: SQIMC-md FMT arm
Procedure: placebo capsule — Oral administration of 30 placebo capsule containing edible pigmented starch
  Arms: Placebo capsule arm

SUMMARY:
This study aims to assess the safety and efficacy of heterologous fecal microbiota transplantation (FMT) by Standardized Quantitative multi-donor Intestinal Microbiota Capsule (SQIMC-md) in mild-moderate ulcerative colitis patients who fail to achieve clinical remission over 4 weeks after full dose 5-Aminosalicylic acid(5-ASA). Intestinal microbiota transplant for FMT will be prepared from multiple healthy donors and prepared by standardized procedure with fixed quantitative dosage. This strategy might offer a novel and safe therapeutic approach for these patients before step up to corticosteroid, immunosuppressant or biologics therapy.

DETAILED DESCRIPTION:
All candidates for mild-moderate ulcerative colitis treated in Dept. Gastroenterology, Tongji Hospital, Tongji Medical College of HUST, the second Xiangya Hospital of central south university and the first affiliated Hospital of Zhengzhou University will be screened for study inclusion and exclusion criteria. All consenting patients will 2:1 randomized into SQIMC-md treatment group or Placebo group. Three dose of SQIMC-md capsule will be orally administrated on day1, day2 and day3. Follow-up will be performed every 4 weeks and last for 12weeks. Full dose of 5-ASA is orally administrated simultaneously during the study. Clinical data and outcome will be collected and documented in electronic case reported form (eCRF).

FMT DONORS:

Potential healthy adult stool donors (between 18 and 28 years of age) will be recruited by the research staff. They will be asked to volunteer for the screening and regularly supply stool samples according to the study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of ulcerative colitis based on clinical symptoms, as well as laboratory and colonoscopic findings, including histopathologic results of the intestinal mucosa.
2. Ulcerative Colitis complete Mayo score range from 4 to 10 [mild-moderate activity] and Mayo endoscopic score ≥2 as assessed within 4 weeks prior to enrollment and clinical symptoms that are at least stable.
3. Patients failed to acquire clinical remission after full dose and adequate course (4 weeks) of 5-ASA or precursors treatment.
4. Patients ≥ 18 and < 70 years of age are eligible for this trial.
5. All patients must sign a written informed consent document. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria:

1. Human immunodeficiency virus (HIV)/acquired immune deficiency syndrome (AIDS) or other severe immunodeficiency
2. Patients with severe prior allergic reaction to food or supplementary material of placebo will be excluded from the protocol.
3. Patients who are pregnant or lactating will be excluded from the protocol.
4. Suspected as CMV or EBV colitis by endoscopic findings and proved by immunohistochemistry and biopsy PCR.
5. Decompensated life-threatening disease including but not restricted to liver cirrhosis (bleeding varices, ascites, encephalopathy or icterus), heart attack, malignancy and so on.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2019-08-30 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate at week 8 after SQIMC-md treatment. | 8 weeks
  Assess efficacy of SQIMC-md FMT treatment with the aid of the Mayo score for Ulcerative Colitis clinical disease severity and response rate at week 8 after SQIMC-md treatment.
  Mayo score (Disease activity index) for Ulcerative Colitis. Total range for complete Mayo score 0-12 (sum from 4 subscales below) and partial Mayo score 0-9 (sum from 1,2 and 4 subscales below):
  Each subscale for mayo score:
  1. Stool frequency: 0-3
  2. Rectal bleeding: 0-3
  3. Mayo endoscopic score: 0-3
  4. Estimation from physician: 0-3
  Clinical response rate is defined as a decrease of ≥ 3 points and at least 30% from baseline in the Mayo score, with an accompanying decrease of ≥ 1 point in the subscore for rectal bleeding or an absolute subscore ≤ 1 for rectal bleeding

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 12 weeks
  safety of SQIMC-md FMT treatment by recording the incidence of adverse events.
clinical response rate at week4 and week12 | week4 and week12
  Assess the efficacy of SQIMC-md FMT by response rate at week4 and week12
the remission rate at week12 | 12 weeks
  the remission rate at week12 with the aid of mayo score or partial Mayo score. Clinical remission rate at week 12 after treatment (clinical remission is defined as a Mayo score of ≤ 2 points and no single score > 1 point
Mean (or median) decrease of fecal calprotectin | 12 weeks
  Assess the efficacy of SQIMC-md FMT measured by the drop of fecal calprotectin.
Mean (or median) change from baseline in Inflammatory Bowel Disease Questionnaire （IBDQ） total score and subscore at week 12 | 12 weeks
  IBDQ includes 32 questions. The questions are grouped into four categories (subscore): Bowel symptoms (B), Systemic symptoms (S), Emotional function (E) and Social function (SF). Response options are consistently presented as seven-point scales (1-7). Total score is defined as the sum of subscore of four categories.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Xiao, Doctoral, Principal Investigator — Tongji Hospital

IPD SHARING:
Plan to Share IPD: Yes
We plan to share at least the ICF and CSR after the trial is ended. The data will be available after we finish the trial and the publication. The sharing of the data is planned to lasted for one year.
Supporting Information: ICF, CSR
Time Frame: The data will be available after we finish the trial and the publication. The sharing of the data is planned to lasted for one year.
Access Criteria: Not decided yet.

REFERENCES:
- [Derived] Huang T, Xu J, Wang M, Pu K, Li L, Zhang H, Liang Y, Sun W, Wang Y. An updated systematic review and meta-analysis of fecal microbiota transplantation for the treatment of ulcerative colitis. Medicine (Baltimore). 2022 Jul 29;101(30):e29790. doi: 10.1097/MD.0000000000029790. PMID 35905229